CLINICAL TRIAL: NCT01847430
Title: Long-term Persistence of Hepatitis B Antibodies and Immune Response to a Challenge Dose of GSK Biologicals' Hepatitis B Virus Vaccine, Engerix™-B Kinder (SKF103860), in 15-16 Years Old Adolescents, Vaccinated in Infancy With Engerix™-B Kinder
Brief Title: Evaluation of the Long-term Persistence of Immunity to Hepatitis B, in Adolescents Vaccinated in Infancy With Engerix™-B Kinder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 116722; 2012-003950-10 (EudraCT Number)
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis B
Keywords: Healthy; Hepatitis B; Adolescents; Engerix™-B Kinder
MeSH Terms: conditions — Hepatitis B

ARMS (1):
- HBV Group (Experimental): Subjects received a single dose of Engerix™-B Kinder vaccine (HBV). The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Engerix™-B Kinder

INTERVENTIONS:
Biological: Engerix™-B Kinder — Single dose administered intramuscularly in the deltoid region of non-dominant arm at Day 0.

SUMMARY:
The purpose of this study is to assess the long-term persistence of immunity to hepatitis B in adolescents aged 15-16 years who were vaccinated with Engerix™-B Kinder in infancy. The study will also assess the immune response to a challenge dose of Engerix™-B Kinder in these subjects.

DETAILED DESCRIPTION:
This MDD has been updated following the Protocol Amendment 1, dated 20 June 2013.

The Protocol was amended because GSK replaced its in-house Enzyme-Linked ImmunoSorbent Assay (ELISA) that was used to measure anti-HBs (antibodies to Hepatitis B surface antigen) antibody concentrations with ChemiLuminescence ImmunoAssay (CLIA).

Additionally, the threshold level of prednisone was modified to reflect the dosage normally prescribed to adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent(s)/guardians who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* A male or female between, and including, 15 and 16 years of age at the time of the vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Written informed assent obtained from the subject in addition to the informed consent signed by the parent(s)/LAR(s).
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Documented evidence of previous vaccination with three consecutive doses of Engerix™-B Kinder in Germany: with the first two doses received by 9 months of age and the third dose received by 18 months of age.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose. For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Previous hepatitis B vaccination since administration of the third dose of Engerix™-B Kinder.
* History of hepatitis B disease.
* Administration of a vaccine not foreseen by the study protocol within the period starting 30 days before study vaccine dose, or planned administration during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥ 37.5°C for oral, axillary or tympanic route, or ≥ 38.0°C on rectal route. The preferred route for recording temperature in this study will be axillary.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the study vaccine dose or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 15 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2013-07-19; Primary Completion 2014-02-21 (Actual); Study Completion 2014-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Germany (10):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Kirchheim, Bavaria
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Neumünster

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Van Der Meeren O, Behre U, Crasta P. Immunity to hepatitis B persists in adolescents 15-16 years of age vaccinated in infancy with three doses of hepatitis B vaccine. Vaccine. 2016 May 23;34(24):2745-9. doi: 10.1016/j.vaccine.2016.04.013. Epub 2016 Apr 16. PMID 27095043
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject from the total number of 303 subjects enrolled did not qualify to start the study due to a protocol violation.
Period: Overall Study
Arm/Group | HBV Group
Started | 302
Completed | 302
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HBV Group
Number analyzed (Participants) | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.3 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 163

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Equal to or Above the Cut Off Value.
Description: The cut-off value was defined as 100 milli-international units per milliliter (mIU/mL).
Time Frame: One month after the challenge dose (Month 1)
Population: The analysis was performed on the according-to-protocol (ATP) cohort of immunogenicity on all evaluable subjects who had received a challenge dose of HBV and for whom data concerning immunogenicity outcome measures were available at the time point after the HBV challenge dose.
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 292
Participants | 265

2. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Equal to or Above the Cut Off Value.
Description: The cut-off values defined were ≥ 6.2 mIU/mL, ≥ 10 mIU/mL and ≥ 100 mIU/mL.
Time Frame: Before (Day 0) and one month after the challenge dose (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 292
Participants
  Day 0 (≥ 6.2 mI/mL) | 208
  Month 1 (≥ 6.2 mI/mL) | 287
  Day 0 (≥ 10 mIU/mL) | 191
  Month 1 (≥ 10 mIU/mL) | 286
  Day 0 (≥ 100 mIU/mL) | 68
  Month 1 (≥ 100 mIU/mL) | 265

3. Secondary Outcome: Antibody Titers Against Hepatitis B Virus
Description: Antibody titers were summarized by geometric mean concentrations (GMCs) with their 95% CIs.
Time Frame: Before (Day 0) and one month (Month 1) after the challenge dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HBV Group
Number analyzed (Participants) | 292
mIU/mL
  Day 0 | 26.5 [21.4 to 32.8]
  Month 1 | 4134.9 [3114.2 to 5490.1]

4. Secondary Outcome: Number of Subjects With an Anamnestic Response to the Challenge Dose in Relation to Their Pre Vaccination Status.
Description: Anamnestic response to the challenge dose was defined as:
  At least (i.e. greater than or equal to ) 4-fold rise in post-vaccination anti-HBs antibody concentrations in subjects seropositive at the pre-vaccination time point Post-vaccination anti-HB antibody concentrations ≥10 mIU/mL in subjects seronegative at the pre-vaccination time point
Time Frame: Prior to vaccination with the challenge dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 291
Participants
  Day 0 < 6.2 mIU/mL: number analyzed (Participants) | 84
  Day 0 < 6.2 mIU/mL | 78
  Day 0 ≥ 6.2 mIU/mL: number analyzed (Participants) | 207
  Day 0 ≥ 6.2 mIU/mL | 204
  Total | 282

5. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as significant pain at rest that prevented normal everyday activities. Grade 3 redness and swelling was greater than 50 millimeters (mm) i.e. >50 mm.
Time Frame: During the 4-day (Days 0-3) follow-up period after the challenge dose
Population: Analysis was performed on the Total Vaccinated cohort which included all subjects who received the challenge dose of HBV vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 302
Participants
  Any Pain | 81
  Grade 3 Pain | 1
  Any Redness | 48
  Grade 3 Redness | 0
  Any Swelling | 16
  Grade 3 Swelling | 0

6. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache and fever [axillary temperature above 37.5 degrees Celsius (°C)]. Gastrointestinal symptoms included nausea, vomiting, diarrhoea and/or abdominal pain. Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = axillary temperature above 39.0°C
Time Frame: During the 4-day (Days 0-3) follow-up period after the challenge dose
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 302
Participants
  Any Fatigue | 84
  Grade 3 Fatigue | 8
  Related Fatigue | 47
  Any Gastrointestinal symptoms | 41
  Grade 3 Gastrointestinal symptoms | 1
  Related Gastrointestinal symptoms | 21
  Any Headache | 67
  Grade 3 Headache | 4
  Related Headache | 41
  Any Fever (≥ 37.5°C) | 7
  Grade 3 Fever (> 39.0°C) | 0
  Related Fever | 4

7. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after the challenge dose
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 302
Participants | 46

8. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs).
Description: Serious adverse event was any untoward medical occurrence that: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (Day 0 to Month 1)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 302
Participants | 2

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: During the entire study period (Day 0 to Month 1), Solicited local and general symptoms: During the 4-day (Days 0-3) follow-up period after the HBV challenge dose.
Arm/Group | HBV Group
Serious Adverse Events (participants affected / at risk) | 2/302
Other Adverse Events (participants affected / at risk) | 169/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HBV Group (N=302)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HBV Group (N=302)
Pain (General disorders) | 81
Swelling (General disorders) | 16
Fatigue (General disorders) | 84
Gastrointestinal symptoms (Gastrointestinal disorders) | 41
Headache (Nervous system disorders) | 67
Redness (General disorders) | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.